CLINICAL TRIAL: NCT00166244
Title: An Open, Prospective, Randomised, Controlled, Multi-Center Study Comparing Fixed Dose vs Concentration Controlled Mycophenolate Mofetil Regimens for de Novo Patients Following Transplantation
Brief Title: Fixed Dose MMF vs Concentration Controlled MMF After Renal Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Dr Teun van Gelder, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDCC
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: De Novo Renal Transplant Recipient.
Keywords: Mycophenolate mofetil; Therapeutic Drug Monitoring; Adult kidney transplantation; Paediatric kidney transplantation
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fixed Dose (Active Comparator): 1 g MMF twice-daily (bid) for adults or 600 mg/m2 bid for paediatric patients. Treatment to be given orally unless it is not possible, in which case it is administered via intravenous (iv) infusion.
  Interventions: Drug: Mycophenolate Mofetil
- Concentration Controlled (Active Comparator): 1 g MMF bid for adults or 600 mg/m2 bid for paediatric patients. Thereafter, MMF doses will be adjusted to MPA AUC0-12 between 30-60mg.h/L based on 3-point abbreviated AUCs (taken at timepoints: 0, 30 min and 120 min always in fasted patients, except for pediatric patients on concomitant tacrolimus) on Days 3 and 10, Week 4, Months 3, 6 and 12 will be performed to determine MPA levels in plasma.
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Mofetil — 1 g for adult patients and 300 mg/m2 for paediatric patients. Fixed dose arm: 1 g twice a day (bid) for adults and 600mg/m2 bid for paediatric patients.
  Concentration controlled arm: initial dose will be 1 g bid for adults and 600mg/m2 bid for paediatric patients. Abbreviated AUCs (taken at timepoints: 0, 30min and 120min in fasted patients) on Days 3 and 10, Week 4, Months 3, 6 and 12 will be performed to determine mycophenolic acid levels in plasma.
  Other Names: CellCept

SUMMARY:
Determine the value of a clinically feasible strategy of therapeutic drug monitoring compared with fixed dosing in de novo MMF treated renal transplant recipients with respect to the incidence of treatment failure.

DETAILED DESCRIPTION:
For treatment with mycophenolate mofetil the contribution of TDM still has to be determined, although circumstantial evidence suggests the measurement of mycophenolic acid plasma concentrations adds to patient management.

A concerted effort to test the hypothesis that TDM will improve outcome in mycophenolate mofetil therapy in a prospective randomised trial is to be made if we want to have a solid base for the continued measurements of mycophenolic acid concentrations in the future. This trial aims to demonstrate the added value of TDM for mycophenolic acid, by comparing fixed dose treatment with concentration controlled mycophenolate mofetil treatment in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients who have completed their second birthday,
* Recipients from living (related or unrelated), cadaveric (non-heart beating or heart beating) donors,
* Single organ recipient (kidney only),
* Women of childbearing potential should have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/ml within 1 week prior to beginning MMF treatment. Effective contraception must be used before beginning therapy, during therapy and for 6 weeks following discontinuation of therapy, even where there has been a history of infertility, unless due to hysterectomy,
* Patients or patient's parent/guardian providing written informed consent,
* Patients co-operative and able to complete all the assessment procedures.

Exclusion Criteria:

* Patients receiving immunosuppressive therapy (except steroid treatment) within the preceding 28 days, except that immunosuppressive medication may be initiated up to 48 hours before transplantation. Furthermore, all patients should receive 1 g [adults] or 600 mg/m2 [paediatric patients] of MMF therapy within 6 hours prior to transplantation,
* PRA > 50% within 6 months prior to enrolment,
* Cold ischaemia time >48 hours,
* History of malignancy (except localised non-melanotic skin cancer) or the presence of any active malignancy at the time of transplant,
* Active peptic ulcer disease,
* Active infection,
* Mandatory intake of prohibited drugs or it is probable that the patient will require treatment with such drugs after transplant,
* Pregnant or lactating females,
* Women of child-bearing potential not willing to use a reliable form of contraception,
* Patient is allergic or intolerant to polysorbate 80 (TWEEN), phenylalanine (aspartame), steroids, MMF, MPA, tacrolimus or cyclosporin,
* Patient or donor with positive tests for HIV or hepatitis B surface antigen,
* Patients with liver cirrhosis or clinical evidence of portal hypertension or other indication of moderate or severe liver disease. (Note: it is strongly recommended that patients with hepatitis C have a liver biopsy performed prior to transplantation),
* Incompatible ABO blood type and/or positive crossmatch,
* Patient has any form of substance abuse, psychiatric disorder or condition, which, in the opinion of the investigator, may invalidate communication with the investigator or with study procedures,
* Patients whose laboratory results reveal severe anaemia (as defined by a haemoglobin value <6 mmol/L [9.7 g/dL] for adults receiving erythropoietin, <4.1 mmol/L [6.6 g/dL] for paediatric patients [regardless of erythropoietin treatment]), leukopenia (as defined by a WBC value of <2500/mm3) or thrombocytopenia (as defined by a platelet count of <75,000/mm3).

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 901 (Actual)
Dates: Start 2003-05; Primary Completion 2005-03 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Treatment failure including the occurrence of the first one of any of the following: biopsy-proven acute rejection, graft loss, death or discontinuation of MMF therapy during the first 12 months following transplantation. | 12 Months

SECONDARY OUTCOMES:
Proportion of patients treated for acute rejection during the first 3, 6, 12 months post-transplantation, | 3, 6 and 12 Months
Time to first acute rejection, | 12 Months
Number of acute rejection episodes per patient in the first year post-transplantation, | 12 Months
Overall treatment outcome at 12 months post-transplantation which is composed of any one of the following: | 12 Months
Graft loss, | 12 Months
Death, | 12 Months
Discontinuation of MMF therapy, | 12 Months
Patient lost to follow-up. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Teun van Gelder, Dr, Principal Investigator — Erasmus Medical Center
Locations (67):
- Australia (7):
  - John Hunter Hospital, New Lambton, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Austria (2):
  - Med. Univ. Klinik, Graz
  - AKH Wien, Vienna
- University Hospitals Leuven, Leuven, Belgium
- Hospital do Rim e Hipertensao, São Paulo, Brazil
- Vancouver General Hospital, Vancouver, British Columbia, Canada
- China (2):
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
- Odense University Hospital, Odense, Denmark
- Surgical Clinic Of Tartu University Clinics, Tartu, Estonia
- France (15):
  - Hopital Pellegrin, C.H.R.de Bordeaux, Bordeaux
  - Hospital du Bocage, Dijon
  - CHU de Grenoble, Grenoble
  - CHU Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hopital Calmette, Lille
  - Hopital Jeanne de Flandres, Lille
  - Centre Hospitalier Regional Universitaire, Limoges
  - CHU Hotel Dieu, Nantes
  - Hopital Necker, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Foch, Suresnes
  - CHU Purpan, Toulouse
  - CHU Rangueil, Toulouse
  - CHU de Nancy-Brabois, Vandœuvre-lès-Nancy
- Germany (6):
  - Universitatsklinikum Charite, Berlin
  - Stadt Kliniken Koln, Cologne
  - Chirurgische Universitätsklinik, Freiburg im Breisgau
  - Universitatsklinikum Heidelberg, Heidelberg
  - University of Heidelberg, Heidelberg
  - University Hospital Wurzburg, Würzburg
- Vilnius University Hospital, Vilnius, Lithuania
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden
  - Erasmus Medical Center Rotterdam, Rotterdam
- Rikshopitalet, Oslo, Norway
- Poland (2):
  - Institute of Transplantology, Medical University of Warsaw, Warsaw
  - Children's Memorial Health Institute, Warsaw
- Spain (14):
  - Hospital Son Dureta, Palma de Mallorca, 07014
  - Hospital Infanta Christa, Badajoz
  - Hospital Del Mar, Barcelona
  - Valle de Hebron, Barcelona
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital de las Nieves, Granada
  - Hospital Ramon Y Cajal, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - La Paz, Madrid
  - Complejo Hospitalario Univeritario de Santiago, Santiago de Compostela
  - Hospital Virgen del Rocio, Seville
  - Hospital Dr. Peset, Valencia
- Sweden (3):
  - University Hospital, Malmo, Malmo
  - Karolinska University Hospital, Huddinge, Stockholm
  - University Hospital A, Uppsala
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (3):
  - Royal Free Hospital, London
  - Guys and St Thomas's Hospital, London
  - St George's Hospital, London
- Venezuela (3):
  - Hospital "Miguel Perez Carreno", Caracas
  - Hospital Universitario de Caracas, Caracas
  - Hospital Universitario de Maracaibo, Maracaibo

REFERENCES:
- [Background] van Gelder T, Hilbrands LB, Vanrenterghem Y, Weimar W, de Fijter JW, Squifflet JP, Hene RJ, Verpooten GA, Navarro MT, Hale MD, Nicholls AJ. A randomized double-blind, multicenter plasma concentration controlled study of the safety and efficacy of oral mycophenolate mofetil for the prevention of acute rejection after kidney transplantation. Transplantation. 1999 Jul 27;68(2):261-6. doi: 10.1097/00007890-199907270-00018. PMID 10440399
- [Result] van Gelder T, Silva HT, de Fijter JW, Budde K, Kuypers D, Tyden G, Lohmus A, Sommerer C, Hartmann A, Le Meur Y, Oellerich M, Holt DW, Tonshoff B, Keown P, Campbell S, Mamelok RD. Comparing mycophenolate mofetil regimens for de novo renal transplant recipients: the fixed-dose concentration-controlled trial. Transplantation. 2008 Oct 27;86(8):1043-51. doi: 10.1097/TP.0b013e318186f98a. PMID 18946341
- [Derived] Hocker B, van Gelder T, Martin-Govantes J, Machado P, Tedesco H, Rubik J, Dehennault M, Garcia Meseguer C, Tonshoff B; FDCC Study Group. Comparison of MMF efficacy and safety in paediatric vs. adult renal transplantation: subgroup analysis of the randomised, multicentre FDCC trial. Nephrol Dial Transplant. 2011 Mar;26(3):1073-9. doi: 10.1093/ndt/gfq450. Epub 2010 Jul 28. PMID 20670958
- [Derived] van Gelder T, Tedesco Silva H, de Fijter JW, Budde K, Kuypers D, Arns W, Soulillou JP, Kanellis J, Zelvys A, Ekberg H, Holzer H, Rostaing L, Mamelok RD. Renal transplant patients at high risk of acute rejection benefit from adequate exposure to mycophenolic acid. Transplantation. 2010 Mar 15;89(5):595-9. doi: 10.1097/TP.0b013e3181ca7d84. PMID 20124953
- [Derived] van Schaik RH, van Agteren M, de Fijter JW, Hartmann A, Schmidt J, Budde K, Kuypers D, Le Meur Y, van der Werf M, Mamelok R, van Gelder T. UGT1A9 -275T>A/-2152C>T polymorphisms correlate with low MPA exposure and acute rejection in MMF/tacrolimus-treated kidney transplant patients. Clin Pharmacol Ther. 2009 Sep;86(3):319-27. doi: 10.1038/clpt.2009.83. Epub 2009 Jun 3. PMID 19494809